CLINICAL TRIAL: NCT07164690
Title: Low-Dose Radiotherapy in Patients With Advanced Esophageal Squamous Cell Carcinoma Resistant to First-Line Chemotherapy Combined With Immunotherapy: a Phase II, Single-arm Study
Brief Title: Low-Dose Radiotherapy in Patients With Advanced Esophageal Squamous Cell Carcinoma Resistant to First-Line Chemotherapy Combined With Immunotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ESOLDRT
Record Dates: First submitted 2025-07-30; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Adenocarcinoma; Radiotherapy
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDRT (Experimental)
  Interventions: Radiation: Low Dose Radiation Therapy

INTERVENTIONS:
Radiation: Low Dose Radiation Therapy — A dose of 2 Gy/1Fx will be delivered to all currently visible lesions. Lesions in different anatomic sites may be irradiated separately, but the entire course must be completed within one week.
  * Esophageal primary tumor management: If the investigator judges there is a risk of fistula or bleeding from the esophageal lesion, palliative radiotherapy at 40-50 Gy may be added.
  * Immunotherapy: The original PD-1/PD-L1 inhibitor regimen will be resumed immediately after LDRT is completed and continued as maintenance therapy.
  * Chemotherapy: At the investigator's discretion, standard second-line chemotherapy per the current CSCO guidelines for esophageal cancer may be administered.

SUMMARY:
Brief Summary

The goal of this single-arm Phase II clinical trial is to learn whether low-dose radiotherapy (LDRT) can restore sensitivity to immunotherapy and prolong disease control in adults with advanced esophageal squamous cell carcinoma who have progressed after first-line chemotherapy combined with PD-1/PD-L1 inhibitors. The main questions it aims to answer are:

* Can LDRT followed by continued immunotherapy increase progression-free survival compared with historical data?
* What is the objective response rate after adding LDRT to ongoing immunotherapy?
* Is LDRT combined with immunotherapy safe in this heavily pre-treated population?

Participants will:

* Receive a single fraction of 2 Gy to every visible metastatic lesion within one week
* Continue their prior PD-1/PD-L1 inhibitor (e.g., camrelizumab, pembrolizumab) after LDRT is completed
* Undergo tumor imaging every 6 weeks for up to one year to monitor response
* Provide optional blood and tissue samples for exploratory biomarker studies

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old;
* ECOG score 0-1;
* Histologically or cytologically confirmed esophageal squamous cell carcinoma that is locally advanced (unresectable) or metastatic (AJCC/TNM 8th edition).
* Progression during or after one prior systemic first-line regimen that contained both a platinum-based chemotherapy and a PD-1/PD-L1 inhibitor (progression must be documented radiologically or clinically). Patients who received neoadjuvant/adjuvant therapy containing a PD-1/PD-L1 inhibitor are considered first-line failures if progression/recurrence occurs during or within 6 months after completion of that therapy.
* At least one measurable lesion per RECIST 1.1 within 4 weeks before enrollment. NOTE: a previously irradiated lesion cannot serve as a target lesion unless clear progression after radiotherapy is documented.
* Life expectancy ≥ 3 months.
* Adequate organ function within 1 week before enrollment:

  * Hematologic: Hb ≥ 80 g/L; WBC ≥ 3.0 × 10⁹/L or ANC ≥ 1.5 × 10⁹/L; platelets ≥ 100 × 10⁹/L.
  * Hepatic: total bilirubin ≤ 1.5 × ULN (direct bilirubin ≤ ULN if total > 1.5 × ULN); ALT/AST ≤ 2.5 × ULN.
  * Renal: serum creatinine < 1.5 × ULN or creatinine clearance ≥ 50 mL/min; BUN ≤ 200 mg/L; albumin ≥ 30 g/L.
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Active autoimmune disease (e.g., inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, vasculitis).
* Symptomatic interstitial lung disease or active infectious/non-infectious pneumonitis.
* Tumor invasion into adjacent organs (aorta or trachea) with high risk of bleeding or fistula; prior esophageal stent placement.
* Other malignancies within the past 2 years (except adequately treated basal-cell carcinoma, cervical carcinoma in situ, etc.).
* Active infection, heart failure, myocardial infarction within 6 months, unstable angina, or uncontrolled arrhythmia.
* Any condition that, in the investigator's opinion, could interfere with study results or increase patient risk.
* Mixed small-cell histology.
* Pregnant or breastfeeding women.
* Congenital or acquired immunodeficiency, HIV infection, prior organ or allogeneic stem-cell transplantation.
* Active HBV, HCV, or tuberculosis infection.
* Prior tumor vaccine or any live vaccine within 4 weeks (inactivated influenza vaccine is allowed).
* Concurrent use of other immunosuppressive agents, chemotherapy, investigational drugs, or chronic corticosteroids.
* Psychiatric illness, substance abuse, or social issues that could compromise compliance.
* Prior intolerance, hypersensitivity, or contraindication to PD-1/PD-L1 inhibitors or chemotherapy components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 1 year

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 year
Objective Response Rate (ORR) | 1 year
Treatment-related adverse event (TRAE) | 1 year

IPD SHARING:
Plan to Share IPD: No